CLINICAL TRIAL: NCT06858371
Title: Effectiveness and Usability of AI-based Chatbots in Improving Depression Literacy, Attitudes Toward Depression, Help-Seeking Intentions, and Confidence in Helping Others: a Randomized Controlled Trial
Brief Title: Testing the Effectiveness of AI Chatbots to Improve Public Knowledge and Attitudes Towards Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Depression Literacy AI Chatbot
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Depression Literacy; Depression Disorders; Stigma of Mental Illness
MeSH Terms: interventions — Training Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AI Depression Education Teacher + AI Depression Patient Simulation Group (Experimental): Participants in this group will interact with two AI-based chatbots, one after the other:
  First Chatbot (Psychoeducation Phase): The first chatbot is designed to provide psychoeducation about depression. Participants will interact with the chatbot to learn key information, such as common symptoms of depression, causes, treatment options, coping strategies, and how to provide emotional support to others experiencing depression. The goal of this phase is to improve participants' understanding of depression and reduce stigma.
  Second Chatbot (Empathy and Support Practice Phase): After completing the psychoeducation phase, participants will interact with a second chatbot simulating a person experiencing depression. This chatbot will simulate real-life conversations, allowing participants to practice empathetic communication, recognize signs of depression, and offer appropriate emotional support.
  Interventions: Behavioral: AI Depression Literacy and Support Training
- Control Group (Active Comparator): Participants in this group will not receive any intervention or access to the Chatbots. Participants will be directed to a depression-related article and a video describing the lived experience of a depression patient.
  Participants in this group will complete the same baseline and post-study assessments as those in the intervention group, which include measures of depression literacy, attitudes toward depression, help-seeking intentions, and confidence in helping others.
  Interventions: Behavioral: Psychoeducation Material Group
- AI Depression Education Teacher Only Group (Experimental): Participants will interact with the AI Depression Education Teacher, an interactive chatbot designed to provide psychoeducation on depression. The chatbot covers topics such as depression symptoms, causes, treatment options, and ways to support individuals experiencing depression. Participants engage in structured conversations and receive real-time feedback to reinforce learning.
  Interventions: Behavioral: AI Depression Literacy Education

INTERVENTIONS:
Behavioral: AI Depression Literacy and Support Training — The intervention consists of two AI-based chatbots designed to enhance depression literacy, reduce stigma, and improve confidence in supporting others with depression.
  AI Depression Education Teacher - This chatbot provides interactive psychoeducation on depression, covering symptoms, causes, treatments, and ways to support others. Participants engage in a structured conversation to enhance their understanding and receive real-time feedback.
  AI Depression Patient Simulation ("Beibei") - Participants interact with a simulated individual experiencing depression to practice empathetic communication and support strategies. Through guided conversations, they learn to recognize depressive symptoms, offer emotional support, and encourage help-seeking.
  This two-phase intervention provides both knowledge and practical experience in a safe, interactive environment. Participants will engage with both chatbots sequentially within a one-hour session.
  Arms: AI Depression Education Teacher + AI Depression Patient Simulation Group
Behavioral: AI Depression Literacy Education — This intervention consists of interaction with an AI chatbot, i.e., AI Depression Education Teacher, which provides interactive psychoeducation on depression, covering symptoms, causes, treatments, and ways to support others.
  Arms: AI Depression Education Teacher Only Group
Behavioral: Psychoeducation Material Group — The intervention contains standard psychoeducation materials about depression. Participants will be directed to:
  A depression-related article - Provides general information about depression, including its symptoms, causes, and treatment options.
  A video describing the lived experience of a depression patient - Shares a personal story to help participants understand the real-life impact of depression.
  Arms: Control Group

SUMMARY:
The purpose of this randomized controlled trial (RCT) is to find out whether using AI Chatbots can help the public better understand depression, reduce negative attitudes towards it, and encourage more people to seek help when needed. The study will also explore whether the Chatbot can help individuals feel more confident in supporting others who might be experiencing depression.

Participants will be randomly assigned to either:

1. AI-PsyTeacher Group: Participants interact with the AI psychology teacher "Liran" to complete three progressive tasks (identifying depression symptoms, learning coping strategies, and understanding prevention). This group assesses the independent role of AI in mental health education.
2. AI-Integrated Intervention Group: Participants first learn with the AI psychology teacher "Liran" and then interact with the AI-simulated depressed patient "Beibei" to complete three tasks (identifying issues, teaching coping strategies, and creating a prevention plan). This group examines the combined effect of AI teaching and patient simulation.
3. Traditional Psychoeducation Group (Control): Participants gain depression-related knowledge by reading traditional educational materials and watching a first-person experience video. This group serves as the control to compare AI interventions.

Primary outcomes include changes in depression literacy, attitudes toward depression, help-seeking intentions, and confidence in helping others. The study aims to determine whether AI-driven interactive learning can improve public understanding and support for mental health.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 65.
2. General population, non-clinical individuals.
3. No history of diagnosed mental disorders or current mental health diagnosis.
4. Ability to complete AI interactions and related tasks via the internet or mobile devices.
5. Native Chinese speakers.
6. Willingness to participate in the study and sign an informed consent form.

Exclusion Criteria:

1. History of mental disorders or self-reported current mental health issues.
2. Currently undergoing psychological counseling.
3. Inability to use mobile or internet devices properly.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Depression Literacy Scale (D-Lit) | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The Depression Literacy Scale is a 22-question survey that assesses a person's depression literacy. The questions are rated on a scale of "true", "false", or "I don't know". Each correct answer is worth one point, with higher scores indicating a higher level of depression literacy.
Depression Literacy Questionnaire | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The Depression Literacy Questionnaire assesses mental health literacy specific to depression. It is a self-developed, 31-item questionnaire designed to assess participants' confidence in providing support to individuals experiencing depression. Each item is rated on a 5-point Likert scale, ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), with higher scores indicating greater depression literacy.
Depression Stigma Scale (DSS) | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The Depression Stigma Scale is designed to measure stigma associated with depression. It has two subscales which measure two different types of stigma: personal and perceived. The Personal Stigma Subscale measures stigma in the respondents own attitudes towards depression by asking them to indicate how strongly they personally agree with nine statements about depression. The Perceived Stigma Subscale measures the respondent's perception about the attitudes of others towards depression by asking them to indicate what they think most other people believe about the same nine statements. Responses to each item are measured on a five-point scale (ranging from zero 'strongly disagree' to four 'strongly agree'). Higher scores indicate higher levels of depression stigma.
Acquisition Questionnaire (AQ-9) | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The Attribution Questionnaire (AQ) is a 9-item self-report assessment tool designed to measure public stigma towards people with mental illnesses. This version assesses emotional reaction and discriminatory responses based on answers to a hypothetical vignette about a man with depression named Xiao Li. Responses assessing stigma towards Xiao Li are in the form of 9 items rated on a Likert scale ranging from 1 (not at all) to 9 (very much).
General Help-Seeking Questionnaire (GHSQ) | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The General Help-Seeking Questionnaire (GHSQ) in this study is an adapted 12-item version designed to fit Chinese cultural contexts. It assesses an individual's intentions to seek help for personal or emotional problems from both formal sources (e.g., mental health professionals, doctors) and informal sources (e.g., family, friends). Each item is rated on a 7-point Likert scale, ranging from 1 ("Extremely Unlikely") to 7 ("Extremely Likely"), with higher scores indicating a greater likelihood of seeking help.
System Usability Scale (SUS) | immediately after the intervention
  The System Usability Scale (SUS) in this study is an adapted 9-item version designed to assess the usability of AI-based chatbots. It evaluates participants' perceptions of the ease of use, effectiveness, efficiency, and overall user experience of the chatbots. The scale uses a 5-point Likert scale, ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), with higher scores indicating better perceived usability. Participants will complete the adapted SUS separately for both the AI Depression Education Teacher and the AI Depression Patient Simulation ("Beibei"). The adapted SUS maintains the core usability assessment principles of the original scale while being tailored for AI-driven conversational agents.
Confidence in Helping Others Scale | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The Confidence in Helping Others Scale is a self-developed, 19-item questionnaire designed to measure participants' confidence in providing support to individuals experiencing mental health issues. Each item is rated on a 5-point Likert scale, ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), with higher scores indicating greater confidence in recognizing depressive symptoms, offering emotional support, and encouraging help-seeking.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ) | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The Patient Health Questionnaire (PHQ-9) consists of 9 items designed to assess the severity of depressive symptoms over the past two weeks. Each item corresponds to one of the nine DSM-5 criteria for major depressive disorder and is rated on a 4-point Likert scale, ranging from 0 ("Not at all") to 3 ("Nearly every day"), with higher scores indicating greater symptom severity.
General Anxiety Disorder (GAD-7) | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report questionnaire used to assess the severity of generalized anxiety symptoms over the past two weeks. Each item corresponds to common symptoms of generalized anxiety disorder (GAD) and is rated on a 4-point Likert scale, ranging from 0 ("Not at all") to 3 ("Nearly every day"), with higher scores indicating greater symptom severity.
Basic Empathy Scale in Adults (BES-A) | pre-intervention, immediately after the intervention, 1-week follow-up, 4-week follow-up, 12-week follow-up
  The Basic Empathy Scale in Adults (BES-A) is a 20-item self-report questionnaire designed to assess an individual's capacity for empathy, including both cognitive empathy (understanding others' emotions) and affective empathy (sharing others' emotions). Each item is rated on a 5-point Likert scale, ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"), with higher scores indicating greater empathy.
Mental Health-Related Behavior Questionnaire | pre-intervention, 4-week follow-up, 12-week follow-up
  This questionnaire is self-conducted and assesses the frequency of various mental health-related behaviors over the past month. Participants rate each behavior based on how often they engaged in it, using a 5-point scale (0 = Never, 4 = More than 4 times per week). The results provide insight into individuals' proactive engagement in mental well-being practices.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university, Beijing, China

IPD SHARING:
Plan to Share IPD: No